CLINICAL TRIAL: NCT01920971
Title: Therapeutic Effects of Monochromatic Infrared Energy Therapy on Patients With Chronic Low Back Pain: A Double-Blind, Randomized, Placebo-Controlled Study
Brief Title: Therapeutic Effects of Monochromatic Infrared Energy Therapy on Patients With Chronic Low Back Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Ru-Lan Hsieh, Associate Professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 102-2314-B-341-001; 102-2314-B-341-001 (Other Grant/Funding Number: National Science Council, Taiwan)
Record Dates: First submitted 2013-08-06; First posted 2013-08-12 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-08

CONDITIONS: Chronic Low Back Pain
Keywords: chronic low back pain; infrared energy; effects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- inferared therapy (Active Comparator): hot pack therapy combined active infrared therapy over the low back (wavelength = 890 nm, radiant power output = 6.24 W, power density = 34.7 milliWatts/cm2 for 40 min, total energy 83.2 J/cm2) followed by 20-min supervised therapeutic exercise, for 3 times per week for a 4-week duration. Patients will be assessed at before treatment and follow-up assessments, including after 2 week of treatment; after 4 weeks of treatment; and 1 and 3 months, respectively, after treatment is terminated.
  Interventions: Radiation: infrared therapy
- placebo infrared therapy (Placebo Comparator): hot pack therapy combined placebo infrared therapy over the low back (wavelength = 890 nm, radiant power output = 6.24 W, power density = 34.7 milliWatts/cm2 for 40 min, total energy 83.2 J/cm2) followed by 20-min supervised therapeutic exercise, for 3 times per week for a 4-week duration. Patients will be assessed at before treatment and follow-up assessments, including after 2 week of treatment; after 4 weeks of treatment; and 1 and 3 months, respectively, after treatment is terminated.
  Interventions: Radiation: infrared therapy

INTERVENTIONS:
Radiation: infrared therapy — wavelength = 890 nm, radiant power output = 6.24 W, power density = 34.7 milliWatts/cm2 for 40 min, total energy 83.2 J/cm2
  Other Names: monochromatic infrared energy therapy

SUMMARY:
To investigate the effects of short-term and medium-term monochromatic infrared energy therapy on patients with chronic low back pain (LBP) according to the International Classification of Functioning, Disability and Health.

DETAILED DESCRIPTION:
Methods：70 participants with chronic LBP will be included. Participants received six 40-min sessions of hot pack therapy combined active or placebo monochromatic infrared energy therapy over the low back (wavelength = 890 nm, radiant power output = 6.24 W, power density = 34.7 milliwatt/cm2 for 40 min, total energy 83.2 J/cm2) followed by 20-min supervised therapeutic exercise, for 3 times per week for a 4-week duration. Patients will be assessed at before treatment and follow-up assessments, including after 2 week of treatment; after 4 weeks of treatment; and 1 and 3 months, respectively, after treatment is terminated.

Main Outcome Measures: Patients will be assessed periodically with pain, Multidimensional Fatigue Inventory, postural stability (using the postural stability evaluation system: Biodex Stability System), and Fear-Avoidance Behavior Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

participants with chronic low back pain

Exclusion Criteria:

1. low back pain accompanied by specific pathological conditions, such as an infection,inflammation, rheumatoid arthritis, fracture, or tumor;
2. a self-reported history of malignancy, vertigo, stroke, or other condition that may impair postural stability;
3. a history of low back surgery with an implant;
4. pregnancy or plans to become pregnant during the course of the study;
5. having received concurrent treatment for low back pain by another health care professional

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-04 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
changes of pain | participants will be evaluated at before treatment, and followed at treatment for 2 and 4 weeks, and 1 and 3 months after treatment
  Participants received six 40-min sessions of hot pack therapy combined active or placebo monochromatic infrared energy therapy over the low back (wavelength = 890 nm, radiant power output = 6.24 W, power density = 34.7 milliWatts/cm2 for 40 min, total energy 83.2 J/cm2) followed by 20-min supervised therapeutic exercise, for 3 times per week for a 4-week duration.

SECONDARY OUTCOMES:
changes of Multidimensional Fatigue Inventory | participants will be evaluated at before treatment, and followed at treatment for 2 and 4 weeks, and 1 and 3 months after treatment
changes of postural stability | participants will be evaluated at before treatment, and followed at treatment for 2 and 4 weeks, and 1 and 3 months after treatment
  using the postural stability evaluation system: Biodex Stability System
changes of fear avoidance behavior | participants will be evaluated at before treatment, and followed at treatment for 2 and 4 weeks, and 1 and 3 months after treatment
  using Fear-Avoidance Behavior Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Lan Hsieh, MD, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan